CLINICAL TRIAL: NCT05811390
Title: Non-surgical Treatment of Periimplantitis - Conventional Hand Instrumentation Versus Air-polishing and Systemic Metronidazole With a 12 Months Follow-up, a Parallel Randomized Controlled Clinical Trial
Brief Title: Non-surgical Treatment of Periimplantitis - Conventional Hand Instrumentation Versus Air-polishing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Periimplantitis treatment
Record Dates: First submitted 2023-02-23; First posted 2023-04-13 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-02

CONDITIONS: Periimplantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- erythritol jet (EMS) (Experimental): An erythritol jet (Perioflow from EMS) will be used to debride the periodontal pockets of oral implants diagnosed with per-implantitis.
  Interventions: Device: erythritol jet
- Manual instrumentation (Active Comparator): An ultrasonic handpiece will be used to debride the periodontal pockets of oral implants diagnosed with per-implantitis.
  Interventions: Device: Manual instrumentation

INTERVENTIONS:
Device: erythritol jet — Use of an erythritol jet in the non-surgical treatment of periimplantitis together with systemic metronidazole
  Arms: erythritol jet (EMS)
Device: Manual instrumentation — Use of manual instrumentation in the non-surgical treatment of periimplantitis together with systemic metronidazole
  Arms: Manual instrumentation

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of ultrasonic instrumentation versus the use of an erythritol jet in the treatment of peri-implantitis.

DETAILED DESCRIPTION:
To carry out this study, the investigators considered a treatment protocol for periimplantitis consisting of 2 phases. The first phase corresponds to the non-surgical treatment of periimplantitis, which can be performed using various techniques. In the present study, it will be carried out using manual instrumentation (with ultrasound and curettes) or with an erythritol jet. In both cases, systemic antibiotic therapy with metronidazole will be performed. The results obtained during the follow-ups will allow the evaluation of the effectiveness of the treatment carried out. If this does not prove to be successful, through an evaluation of clinical and radiographic criteria, patients will be advised to undergo a second phase of treatment, in this case a surgical treatment of peri-implantitis, but which will no longer be part of the interventions carried out and documented in this study. Patients for whom the unsatisfactory treatment was considered effective will be allocated to a periimplant support treatment program, which means that they will be advised to carry out maintenance consultations at the FMDUP clinic with a specific and individualized periodicity in order to maintain the health of the periimplant tissues and the remaining oral cavity. The study will be carried out by the students of the Specialization in Periodontology and Oral Implantology 2021-2024 of the Faculty of Dental Medicine of the University of Porto (FMDUP).

ELIGIBILITY:
Inclusion Criteria:

* At least 1 osseointegrated implant diagnosed with peri-implantitis (according to the new Classification of Periodontal and Peri-implant Diseases and Conditions) and rehabilitated with screw-retained crown
* Patients of legal age (≥18 years old)

Exclusion Criteria:

* Uncontrolled systemic pathologies, namely diabetes mellitus (HbA1c > 7% or >53 mmol/mol)
* Pregnant or lactating patients
* Severe smoking (>20 cigarettes/day)
* Systemic pathologies, medication or treatments that cause alterations in bone metabolism (for example: osteoporosis, bisphosphonates, radiotherapy of the head and neck)
* Patients who missed study control visits
* Patients who have received systemic antibiotic therapy in the last 2 months
* Patients with allergies to any of the components used in the study, namely to erythritol
* Implants that have previously undergone surgical treatment for peri-implantitis
* Implants with bone loss greater than 2/3 of their length and/or mobility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Change in probing pocket depth | 0, 3, 6, 12 months
  The distance measured from the base of the sulcus or pocket to the free gingival margin at six points per implant (measured in millimetres).

SECONDARY OUTCOMES:
PROMS | 0 months
  Patient reported outcomes reported on a visual analog scale from 0 (no pain) to 10 (maximum pain).
Change in alveolar bone level | 0,12 months
  Radiographically measured alveolar bone level from the alveolar crest to the implant's neck, mesially and distally (measured in millimetres).
Change in gingival recession | 0, 3, 6, 12 months
  Gingival recession measured at six points per implant with a periodontal probe, from the cementum-enamel junction to the bottom of the probable pocket (measured in millimetres).
Bleeding on probing | 0, 3, 6, 12 months
  Bleeding on probing (in percentage) assessed 30 seconds after probing, through a dichotomous scoring system used at six sites per implant using one (1) and zero (0) for presence or absence, respectively.
Implant survival rate | 0, 12 months
  Percentage of implants that survived after 1 year follow-up (implants that remain in the patient's mouth after 1 year).

CONTACTS AND LOCATIONS:
Overall Officials: Ana Isabel Moreira, Principal Investigator — Faculdade de Medicina Dentária da Universidade do Porto
Locations (1):
- Faculty of Dentistry at the University of OPorto, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No